CLINICAL TRIAL: NCT07238751
Title: Effects of Bowen Technique With Retro-walking on Hamstring Flexibility in Knee Osteoarthritis Patients
Brief Title: Bowen Technique With Retro-walking on Hamstring Flexibility in Knee Osteoarthritis
Acronym: A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aqsa Butt
Record Dates: First submitted 2025-09-25; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Hamstring tightness; Bowen technique; Retro-walking
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowen technique with Retro-walking (Other): Bowen technique with Retro-walking
  Interventions: Other: Bowen technique with Retro-walking
- Conventional PT (Other): Conventional PT
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Other: Bowen technique with Retro-walking — In initially step the patient in prone position and therapist approach on the same side of the treatment limb. Use the thumb by applying the pressure on the lateral side of the target muscle. The treatment sequence will begin with thumb gradually involve the finger. a single treatment consists of a series of specific sequences of these moves with frequent pauses 2 to 5 minutes to allow time for the body to respond. Treatment session duration 15-20 minutes occur 3 days per week, for 4 weeks. Week 1(retro-walking on flat surface for 5 minutes) week 2(retro walking on flat surface for 7 minutes) week 3(retro-walking on flat surface for 10 minutes) week 4 (retro-walking on flat surface for 15 minutes) .Conventional PT including 1- hot pack 2-isometric quadriceps exercise(1 set of 10 reps twice a day)2-SLR stretch (1set of 10 reps twice a day)4-isometric hip adduction exercise( 1 set of 10 reps twice a day)5-Terminal knee extension( 1 set of 10 reps twice a day) total duration is 3 sessions
  Arms: Bowen technique with Retro-walking
Other: Conventional Treatment — Conventional PT including 1-. Hot pack 2- isometric quadriceps exercise (1 set of 10 reps twice a day) 3-SLR Stretch (1set of 10 reps twice a day) 4 -isometric hip adduction exercise (1 set of 10 reps twice a day) 5-Terminal knee extension (1 set of 10 reps twice a day) Total duration is 3 sessions per week for 4 consecutive weeks.
  Arms: Conventional PT

SUMMARY:
The aim of this randomized controlled trial is to find the effects of Bowen technique with retro-walking on hamstring flexibility, pain, dynamic mobility and knee related disability in knee Osteoarthritis patients

DETAILED DESCRIPTION:
The term osteoarthritis is also known as degenerative joint disease because of wear and tear process occur in articular cartilage. OA affect the joints, the tissue surrounding the joint and other connective tissue. The symptoms of knee OA is most common seen in obese and aged individuals. There are three compartment that affected in knee OA include medial, lateral and patellofemoral joint. The OA takes 10 to 15 years to develop. The pathophysiology of the OA is still under investigation. Traditionally it was considered that it was due to aging factor because wear and tear process occur in articular surfaces.

But now it's considered there are multiple factors that involve in the origin of OA include biomechanical and inflammatory factors. Knee OA is influenced by family history, age, obesity, joint shape, genu valgus and varum and inflammation by metabolic syndrome. In radiological findings wo notice that bony osteophytes, damaging of articular cartilage, sclerosis of the subchondral bone seen, and it's become severe later. Knee OA may be modified or may be unmodified. In unmodifiable include genetically or congenital. But in modifiable is excessive weight. In Modern treatment we focus on improve the function limitation and quality of life which we can improve by physiotherapy Several muscles are involved in the support of knee. The 2 major muscle groups quadriceps and hamstrings are involved in the movement and stability of the knee joint. The quadriceps and hamstrings provide the knee stability in frontal plane. In knee OA pathogenesis important muscle imbalance arise from quadriceps group of muscles or hamstring group of muscles weakness, which is usually assessed by quadriceps hamstrings ratio(Q:H). In knee OA medial compartment of tibiofemoral joint is mostly involved.

Bowen technique helps in restore the fascia disturbances and muscle imbalances. During the application of the Bowen technique, it stimulates the brain ascending neural impulses to allow the fascia changes this mechanism is called fascia plasticity.) Bowen therapy works on our body nervous system by stimulating the parasympathetic nervous system and encourage the state of relaxation and healing. Bowen moves are applied on the muscle's origin, insertion, or belly of muscles where Golgi receptors are located. Bowen therapy improves body ability to function at a cellular level.

Backward walking increases the coordination because during backward walking isometric and concentric activity both are occurred. The backward walking mechanism is different from the forward walking, in backward walking toes contact the ground first and the heel is lifted off the ground in early stance. Retro walking can minimize the burden on the joint and increase the muscle length in normal healthy individuals.

This study aims to find the effects of Bowen technique with retro-walking on hamstring flexibility, pain, dynamic mobility and knee related disability in knee Osteoarthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-60 years
* Both gender: male and female
* Less than 80-degree hip flexion angle on passive SLR, Active knee extension greater than 20 indicates hamstring muscle tightness
* Kellgren and Lawrence classification (stage I and stage II)
* Bilateral hamstring tightness
* Visual analogue scale value greater than 3
* Pain duration more than 3 months

Exclusion Criteria:

* Meniscal injury or ligamentous injury
* Muscle/tendon injuries of hamstring
* Spinal Injuries and any other co- morbidity
* Any surgery, infection, trauma, pregnancy, fracture and fall
* Involvement in regular flexibility yoga program
* Patient with intra articular steroidal therapy with in last 6 months
* Patient involvement in another intervention study
* Malignancy
* Pregnancy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue scale VAS | 4 weeks
  The VAS is psychomotor response scales to investigate a unidimensional measure of pain intensity. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Active knee extension test | 4 weeks
  Active knee extension will use to access the flexibility of the hamstring muscle. Ask the patient to lay down in spine position while flexing the hip 90-degree, other leg down with couch and leg to be test with both hands. The goniometer will place on knee and ask the patient to extend the knee holding hip flex 90 degree
SLR | 4 weeks
  A goniometer will be used to measure the range of hip flexion on passive SLR and range less than 80 degree indicate that the hamstring muscle tightness
Timed Up and Go (TUG) Test | 4 weeks
  The TUG test measures the time taken by a participant to stand up from a standard chair, walk a distance of 3 meters, turn around, walk back to the chair, and sit down. It assesses dynamic balance and functional performance.
Knee injury and osteoarthritis score | 4 weeks
  In KOOS include 42 items in five subscales to check different categories i.e. pain (9 items), symptoms (7 items), functions in the activity of daily living (ADLs) (17) items), sports and recreational activities (5 items), and quality of life (4 items).

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Shaafi international hospital,ISLAMABAD, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No